CLINICAL TRIAL: NCT05363475
Title: Implementation and Evaluation of a Continuous Bedside Pressure Mapping System in Multiple Patient Care Settings
Brief Title: Implementation and Evaluation of CBPM Technology
Acronym: CBPM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Barry Baylis (Other)
Collaborators: XSENSOR Technology Corporation (Unknown)
Responsible Party: Sponsor-Investigator, Barry Baylis, Clinical Associate Professor, University of Calgary
Organization: University of Calgary (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REB22-0239
Record Dates: First submitted 2022-05-02; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Pressure Injury; Surgical Wound
MeSH Terms: conditions — Pressure Ulcer; Surgical Wound

STUDY DESIGN:
Intervention Model Description: Prospective cohort with comparison to retrospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prospective (Experimental): Participants will be monitored by the ForeSite Intelligent Surface system for 2-3 weeks.
  Interventions: Device: ForeSite Intelligent Surface

INTERVENTIONS:
Device: ForeSite Intelligent Surface — The ForeSite IS is a continuous bedside pressure mapping system with machine learning and artificial intelligence (ML/AI). It consists of an overlay with over 1500 undetectable integrated sensors and a medical-grade bedside touchscreen monitor. The monitor displays a real-time coloured body pressure image, a turn timer, and a history of previous turns. The ML/AI software tracks 17 body locations and the patient's body position. The system has a centralized dashboard that shows the pressure injury risk and turn history, which can be transmitted to the nursing station. In addition, data is stored in an Amazon Web Services (AWS) secured cloud database, enabling access to individual reports on turn history and compliance and pressure exposure. Data is stored as both, raw pressure data files and real time event information on pressure exposure and turn data.
  Other Names: ForeSite IS

SUMMARY:
Background & Rationale: Pressure injuries are costly to treat and are prevalent in about 26% of patients across all healthcare settings in Canada. Wounds Canada has developed recommendations for prevention and management to tackle this problem that include pressure injury risk assessment, pressure relief surfaces, nutrition, wound monitoring, and wound care. Continuous bedside pressure mapping (CBPM) technology can assist with effective repositioning of patients to prevent pressure injuries. The ForeSite Intelligent Surface system (ForeSite IS) is a CBPM technology that uses machine learning and artificial intelligent software for more intuitive repositioning of patients. Various studies have shown the technology to be effective in reducing pressure injuries and providing adequate pressure redistribution for patients with a PI flap reconstruction. Furthermore, some studies have indicated the device's cost savings, but there are no known publications on cost-effectiveness. Despite the few studies evaluating CBPM technology, few have implemented it in nursing care. Particularly in Canada, there are no guidelines for incorporating CBPM technology into pressure injury prevention care plans or post-surgical recovery in any healthcare setting.

Research Question and Objectives: In this study we will be piloting the ForeSite IS system in long-term care, acute care, plastic surgery and trauma patients to further identify the benefits of utilizing the device and evaluate its implementation. The primary objectives are:

1. To determine if the ForeSite IS system can be incorporated in improving quality of care for at risk patients by providing continuous skin exposure monitoring
2. To determine if the ForeSite IS system can provide evidence of skin breakdown to reduce the incidence and risk of PIs
3. To determine if the ForeSite IS system can assist with offloading of pressure to improve healing of post-surgical patients

The secondary objectives are:

1. To determine if the device improves nursing workflow and productivity
2. To determine the cost-effectiveness of using the ForeSite IS system

Methods: The ForeSite IS system will be piloted in long-term care and acute care for six months. The researchers will identify patients with nursing staff and get permission to approach them. Once permitted, they will explain the study and obtain written consent from patients who agree to participate. Nursing staff will be responsible for setting up and removing the device from the patient's bed. For the first 48 hours of monitoring with the device, no visual feedback (blinded period) will be provided to the nursing staff to collect interface pressure and patient repositioning data on current care practices. Nursing staff will then have another 48 hours to use the visual feedback from the device and acclimatize to the device (acclimatization period). Afterwards, nursing staff will use the visual feedback for the remainder of the patient's two to three weeks of monitoring (active period), depending on the clinical setting. Nurses will continue with routine skin assessments throughout the entire monitoring with additional skin assessments if prompted by the visual feedback during the active period. Interface pressure and patient repositioning in the first 48-hour blinded period will be compared to the monitoring period after the 48-hour acclimatization period. After implementation of the pilot, clinical outcomes will be compared to clinical outcomes of a six-month period prior to the pilot.

Pre-implementation focus groups/interviews will be conducted with nursing staff to help each clinical setting develop a protocol for using the ForeSite IS system and develop strategies for implementation. Post-implementation focus groups/interviews will be conducted one to two months after implementation of the system to understand the system's barriers, facilitators, and sustainability aspects.

ELIGIBILITY:
For evidence of skin breakdown:

Inclusion Criteria:

* adults that require assistance with bed mobility or are entirely dependent for bed mobility based on de Morton Mobility Index, ability to provide consent or have a legal representative to provide consent on their behalf, expected length of stay is more than 14 days

Exclusion Criteria:

* near end of life, have a planned admission to another unit, their clinical care would be negatively impacted if turned or repositioned, increased mobility

For post-surgical repair:

Inclusion Criteria:

* adults, flap repair where the donor or recipient site is on the posterior side of the patient, or trauma patients with a surgical procedure on the posterior side of the patient, ability to provide consent or have a legal representative to provide consent on their behalf, partially or entirely dependent on mobility for the first 14-21 days post-surgery, ALOS is over 14 days

Exclusion Criteria:

* a patient has complications that result in near end of life with death imminent, the patient becomes more mobile (e.g., can sit up from supine without assistance or can roll to the side without assistance) in less than 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Incorporating the ForeSite IS in nursing care | 2-3 weeks during monitoring
  Compliance of repositioning patients according to the system and recommended turning regimen by clinician, and feedback from nursing staff during focus groups
Providing evidence of skin breakdown | 2 weeks during monitoring
  Incidence of pressure injuries and skin assessments correlated to average interface pressure, average pressure exposure and peak pressure
Improves healing of surgical wounds | 2-3 weeks during monitoring
  Skin and surgical site infections correlated to average interface pressure, average pressure exposure and peak pressure

SECONDARY OUTCOMES:
Improving nursing workflow | 2-3 weeks
  rate of repositioning per day, average exposure time between repositions and duration of body positions
Cost-effectiveness | 6 months
  cost of care per quality adjusted life year

CONTACTS AND LOCATIONS:
Overall Officials: Barry W Baylis, MD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No